CLINICAL TRIAL: NCT05460208
Title: Hypocholesterolemic and Cardioprotective Clinical Evaluation of a Spreadable Cream Prepared With Virgin Olive Oil Enriched in Phytosterols and Bioactive Compounds From Olives in Children and Adolescents
Brief Title: Hypocholesterolemic Effect of a Phytosterol-enriched Spreadable Cream Prepared With Virgin Olive Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government); Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Principal Investigator, María Dolores Mesa García, Professor, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MEDKIDS-Chol; IDI-20190983 (Other Grant/Funding Number: Centro de Transferencia Tecnológica - UGR)
Record Dates: First submitted 2022-03-07; First posted 2022-07-15 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Hypercholesterolemia
Keywords: Virgin olive oil; Plant Sterols; Hypercholesterolemic children; Olive oil polyphenols
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enriched spread (Experimental): Children between 20-40 kg will receive a dose of 15 g of the spread (1.2 g/d of plant sterols: 0.06-0.03 g/kg of weight/d) and those with a weight between 40-60 kg will receive two doses of 15 g of the spread (2.4 g/d of plant sterols: 0.06-0.04 g/kg of weight/d)
  Interventions: Dietary Supplement: Enriched spread
- Control spread (Placebo Comparator): Children between 20-40 kg will receive a dose of 15 g of the spread (1.2 g/d of plant sterols: 0.06-0.03 g/kg of weight/d) and those with a weight between 40-60 kg will receive two doses of 15 g of the spread (2.4 g/d of plant sterols: 0.06-0.04 g/kg of weight/d)
  Interventions: Dietary Supplement: Control spread

INTERVENTIONS:
Dietary Supplement: Enriched spread — The experimental spread is made with a base made with 90% extra virgin olive oil to which plant sterols are added.
  Arms: Enriched spread
Dietary Supplement: Control spread — The control spread will be the same base spread made with extra virgin olive oil without the added plant sterols.
  Arms: Control spread

SUMMARY:
This study aims to evaluate the effect of the enriched extra virgin olive oil spread in plant sterols from the olive itself and demonstrate its effect anticholesterolemic and cardioprotective in children and adolescents with hypercholesterolemia.

DETAILED DESCRIPTION:
A clinical study of nutritional intervention, randomized with double blind, adjusted by randomization blocks that consider age and sex, and crossover of 2 months duration each period, with 1-month washout period, in 50 subjects (25 per randomization group). The study will be carried out in the Reina Sofía Universitary Hospital of Córdoba, as well as at the Institute of Nutrition and Food Technology of the University of Granada.

The effects of the enriched spread in patients on the lipid profile will be evaluated plasma and its action on biomarkers of cardiovascular risk and on the microbiota intestinal depending on the specific genotype of each subject. In addition, the presence of minor olive oil compounds present in plasma (metabolomic analysis). In this way, at the end of the project, scientific information will be available contrasted on the enriched product and its effects on cardiovascular protection, in addition to its palatability and acceptance.

The main objective is to evaluate the effect of the enriched extra virgin olive oil spread in plant sterols from the olive itself and demonstrate its effect anticholesterolemic and cardioprotective in children and adolescents with hypercholesterolemia.

As specific objectives will be determined:

* To evaluate the effect of the enriched spread on the plasmatic concentrations of total cholesterol, LDLc and other parameters of the lipid profile
* To evaluate the effect of the enriched spread on the oxidative status of LDL plasmatic
* To evaluate the effect of the enriched spread on the antioxidant defense system
* To evaluate the effect of the enriched spread on biomarkers of cardiovascular risk, including inflammatory and endothelial damage markers
* To evaluate the effect of the enriched spread on the intestinal microbiota.
* To evaluate the effect of the enriched spread on the metabolomic changes in plasma.
* To analyze the specific genotype of each volunteer

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 18 years
* Familial hypercholesterolemia
* Acceptance to participate by signing the informed consent

Exclusion Criteria:

* Children under 6 years of age
* Absence of hypercholesterolemia
* Children who receive some type of medication to control hypercholesterolemia, blood pressure, levels of glucose or dyslipidemia or any probiotic, which have invalid data for the variables of the present study
* Not to sign the informed consent.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Hypercholesterolemia | Month 0; Month 2; Month 3; Month 5
  Assessing changes of plasma lipids levels from the baseline to the end of each treatment. The serum concentrations of total cholesterol (mg/dL), triglycerides (TG, (mg/dL)), high-density lipoprotein cholesterol (HDLc, (mg/dL)), and low-density lipoprotein cholesterol (LDLc, (mg/dL)), apolipoprotein A1 (Apo-A1, (mg/dL)) and apolipoprotein B (Apo-B, (mg/dL)) will be analyzed by spectrophotometry.

SECONDARY OUTCOMES:
Body composition | Month 0; Month 2; Month 3; Month 5
  Assessing changes of body composition from the baseline to the end of each treatment. To obtain data on body composition, fat mass (kg), lean mass (kg) and total body water (kg) will be measured via bioimpedance technology using TANITA MC-780MA (Tokyo, Japan).
Body composition percentages | Month 0; Month 2; Month 3; Month 5
  Assessing changes of body composition percentages from the baseline to the end of each treatment. To obtain data on body composition, fat mass (percent), lean mass (percent) and total body water (percent) will be measured via bioimpedance technology using TANITA MC-780MA (Tokyo, Japan).
Systolic blood pressure | Month 0; Month 2; Month 3; Month 5
  Assessing changes of Systolic Blood Pressure from the baseline to the end of each treatment.
Diastolic blood pressure | Month 0; Month 2; Month 3; Month 5
  Assessing changes of Diastolic Blood Pressure from the baseline to the end of each treatment.
Oxidation biomarkers | Month 0; Month 2; Month 3; Month 5
  Assessing changes of oxidized LDL from the baseline to the end of each treatment, by using an ELISA kit
Enzymatic antioxidant status | Month 0; Month 2; Month 3; Month 5
  Assessing changes on erythrocyte antioxidant enzymes (catalase, superoxide dismutase, glutathione peroxidase and glutathione reductase) from the baseline to the end of each treatment, by using spectrophotometric kits.
Non-enzymatic antioxidant status | Month 0; Month 2; Month 3; Month 5
  Assessing changes on plasma liposoluble antioxidants (retinol, beta-carotene and Q-coenzyme) from the baseline to the end of each treatment, by HPLC.
Endothelial function status | Month 0; Month 2; Month 3; Month 5
  Assessing changes on plasma endothelin-1 from the baseline to the end of each treatment, by using an ELISA kit.
Endothelial damage | Month 0; Month 2; Month 3; Month 5
  Assessing changes on plasma VCAM , ICAM-1, E-selectin and mielopeoxidasa from the baseline to the end of each treatment, by Luminex xMAP technology.
Fecal microbiome | Month 0; Month 2; Month 3; Month 5
  Assessing changes of fecal microbiome profile from the baseline to the end of each treatment. Stool DNA will be isolated with the QIAamp DNA stool mimi kit. Amplification of variable region V3-V1 of 16S gen will be sequenced using the Illunina Next Generation Sequencing MiSeg.
Plasma metabolomic analysis | Month 0; Month 2; Month 3; Month 5
  A liquid chromatography platform coupled to a spectrophotometer will be used mass (LC/MS) to determine plasma metabolic profiles by targeted analyses from the baseline to the end of each treatment.
Urine metabolomic analysis | Month 0; Month 2; Month 3; Month 5
  A liquid chromatography platform coupled to a spectrophotometer will be used mass (LC/MS) to determine urine metabolic profiles by targeted analyses from the baseline to the end of each treatment.

CONTACTS AND LOCATIONS:
Overall Officials: MARÍA DOLORES MESA GARCÍA, Principal Investigator — Universidad de Granada
Locations (2):
- Spain (2):
  - Hospital Universitario Reina Sofia de Córdoba, Córdoba
  - Universidad de Granada, Granada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Perez P, Vazquez-Aguilar A, Sanchez-Rodriguez E, Jurado-Castro JM, Pastor-Villaescusa B, Gil-Campos M, Rangel-Huerta OD, Gil A, Aguilera CM, Mesa MD, Rocchetti G, Lucini L. Chemometrics-guided plasma lipidomics insights underlying the decrease of plasma total cholesterol and LDLc in children with hypercholesterolemia following habitual intake of an EVOO-based phytosterols-enriched spreadable cream. Metabolomics. 2025 Nov 15;21(6):169. doi: 10.1007/s11306-025-02368-3. PMID 41241688